CLINICAL TRIAL: NCT06093139
Title: Monocentric Crossover Study to Assess the Tolerability and the Efficacy of a Mix of Probiotic Strains Doses vs Placebo in Athletes Performance
Brief Title: Efficacy of a Mix of Probiotics in Athletes Performance
Acronym: GIU-PPA-0420
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giuliani S.p.A (Industry)
Collaborators: FitBiomics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: GIU-PPA-0420
Record Dates: First submitted 2023-05-21; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-05

CONDITIONS: Healthy
Keywords: athletes; probiotics; performance
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Probiotic capsule (composition same as described above - L. acidophilus FB0012, L. plantarum FB0015, and L. rhamnosus FB0047 encapsulated in acid-resistant capsules alongside additional potato starch as a filler).
  Interventions: Dietary Supplement: Probiotic capsule
- Placebo (Placebo Comparator): Placebo capsule (placebo consisted of the same capsules filled with potato starch)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic capsule — probiotic capsule (composition same as described above - L. acidophilus FB0012, L. plantarum FB0015, and L. rhamnosus FB0047 encapsulated in acid-resistant capsules
  Other Names: L. acidophilus FB0012, L. plantarum FB0015, and L. rhamnosus FB0047 encapsulated in acid-resistant capsules
  Arms: Active
Dietary Supplement: Placebo — placebo consisted of the same capsules filled with potato starch
  Arms: Placebo

SUMMARY:
Monocentric Crossover Study to Assess the Tolerability and the Efficacy of a Mix of Probiotic Strains Doses vs Placebo in Athletes Performance

This study will intend:

- To assess the tolerability and the efficacy of a food supplements into improving performance in a panel of athletes after repeated use for 4 consecutive weeks, under the normal conditions of use, compared to a placebo.

DETAILED DESCRIPTION:
The present study aimed at assessing the tolerability and the efficacy of a food supplements probiotics-based (L. acidophilus FB0012, L. plantarum FB0015, and L. rhamnosus FB0047 encapsulated in acid-resistant capsules) into improving performance in a panel of athletes after repeated use for 4 consecutive weeks, under the normal conditions of use, compared to a placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female athletes18-45 years old (included).
2. Subjects accepting to follow the instruction received by the investigator and disposable and able to return to the study centre at the established times.
3. Subjects accepting to not receive any drugs/cosmetics treatment able to interfere with the study results.
4. No participation in a similar study actually or during the previous 6 months.
5. Subjects accepting to sign the Informed consent form.

Exclusion Criteria:

* 1. Known sensitivity to any compound of the Investigational product. 2. Pregnant or breast feeding females or planning a pregnancy. 3. Serious intercurrent infection or other active disease up to three months prior to study entry.

  4. History of concurrent malignancy. 5. History of significant alcohol or drug abuse. 6. Significant psycho-social or psychiatric disorders that may impair the subject's ability to meet the study requirements.

  7. Significant concurrent medical disorders that may impair the subject's ability to participate over the whole one year of the study.

  8. Any other medical condition which in the Investigator's opinion would prevent the subject from participating in the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of physical parameters: soreness | at T1 (12 weeks with placebo) and T1 (12 week with ACTIVE)
  Change of Soreness (measured by a 5-point scale) between T1 and T2
Evaluation of physical parameters: fatigue | at T1 (12 weeks with placebo) and T1 (12 week with ACTIVE)
  Change of Fatigue (measured by a 5-point scale) between T1 and T2
Evaluation of physical parameters: energy | at T1 (12 weeks with placebo) and T1 (12 week with ACTIVE)
  Change of Energy (measured by a 5-point scale) between T1 and T2between T1 and T2
Evaluation of physical parameters:Sleep quality | at T1 (12 weeks with placebo) and T1 (12 week with ACTIVE)
  Change of Sleep quality (evaluated by Sleep Quality Scale (SQS)) between T1 and T2between T1 and T2
Evaluation of physical parameters:Digestive symptoms | at T1 (12 weeks with placebo) and T1 (12 week with ACTIVE)
  Change of the frequency of four individual digestive symptoms (abdominal pain/discomfort, bloating, flatulence/passage of gas and borborygmi/rumbling stomach) will be evaluated with five-point Likert scales that range from 0 (never) to 4 (every day of the week), between T1 and T2
Gut microbiota analysis ON FECAL SAMPLE by mean of 16S and metagenomic shotgun sequencing | at baseline (T0)
  16S and metagenomic shotgun sequencing
Gut microbiota analysis ON FECAL SAMPLE by mean of 16S and metagenomic shotgun sequencing | at T1 (12 weeks with placebo) a
  16S and metagenomic shotgun sequencing
Gut microbiota analysis ON FECAL SAMPLE by mean of 16S and metagenomic shotgun sequencing | at T1 (12 week with ACTIVE)
  16S and metagenomic shotgun sequencing
Microbial dysbiosis ON URINE SAMPLES by mean of liquid chromatography- surface-activated chemical-ionization-electrospray ionization (LC/SASI-MS) and tandem mass spectrometry (MS/MS) | at baseline (T0),
  By mean of liquid chromatography bacteria that potentially could cause dysbiosis by analyzing the profile of urine's metabolites and combining the results in the SANIST platform which predicts the intestinal dysbiosis based on the antagonist and pathogen bacteria pharmacological activity
Microbial dysbiosis ON URINE SAMPLES by mean of liquid chromatography- surface-activated chemical-ionization-electrospray ionization (LC/SASI-MS) and tandem mass spectrometry (MS/MS) | at T1 (12 weeks with placebo)
  By mean of liquid chromatography bacteria that potentially could cause dysbiosis by analyzing the profile of urine's metabolites and combining the results in the SANIST platform which predicts the intestinal dysbiosis based on the antagonist and pathogen bacteria pharmacological activity
Microbial dysbiosis ON URINE SAMPLES by mean of liquid chromatography- surface-activated chemical-ionization-electrospray ionization (LC/SASI-MS) and tandem mass spectrometry (MS/MS) | T1 (12 week with ACTIVE)
  By mean of liquid chromatography bacteria that potentially could cause dysbiosis by analyzing the profile of urine's metabolites and combining the results in the SANIST platform which predicts the intestinal dysbiosis based on the antagonist and pathogen bacteria pharmacological activity

CONTACTS AND LOCATIONS:
Overall Officials: DANIELA PINTO, Study Chair — Giuliani S.p.A
Locations (1):
- Centro Sportivo Parma Football, Collecchio, Parma, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/39/NCT06093139/ICF_000.pdf